CLINICAL TRIAL: NCT06864689
Title: Leveraging Video Logs as a Bridge to Pre-exposure Prophylaxis (PrEP) With Tailored Messaging to Black Women and Their Healthcare Providers in Texas.
Acronym: PrEP
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-0363; 1R34MH136826-01 (NIH)
Record Dates: First submitted 2025-02-13; First posted 2025-03-07 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: HIV Prevention
Keywords: Minoritized population; Video logs; PrEP; Health communication; Behavioral intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): Participants will watch a health-informed video-log series and complete a second survey (post-test). The post-test will assess the same variables previously assessed in the pre-test.
  Interventions: Behavioral: Video-log (vlog) series with videos tailored to cisgender Black women or to healthcare providers
- Standard of Care (No Intervention): Participant will receive SOC and complete the post-test.

INTERVENTIONS:
Behavioral: Video-log (vlog) series with videos tailored to cisgender Black women or to healthcare providers — This intervention is a video-log (vlog) series based health communication intervention that will be disseminated through community health centers (CHCs) and social media to increase willingness for and use of PrEP among cisgender Black women and to increase willingness to prescribe and refer PrEP among healthcare providers.
  Arms: Intervention

SUMMARY:
The primary objective of this R34 proposal is to increase willingness for PrEP initiation and PrEP initiation among Black Women (BW) and increase willingness to prescribe/refer pre-exposure prophylaxis (PrEP) to CBW among healthcare providers (HCPs) in Houston/Harris County, a high priority Ending the HIV Epidemic (EHE) jurisdiction.

DETAILED DESCRIPTION:
The primary objective of this R34 proposal is to increase willingness for pre-exposure prophylaxis (PrEP) initiation and actual PrEP initiation among BW, increase willingness to prescribe/refer PrEP to BW among HCPs in Houston/Harris County, a high-priority End the HIV Epidemic (EHE) jurisdiction. The investigator hypothesizes that a video-log (vlog) series-based health communication intervention disseminated through community health centers (CHCs) and social media will increase willingness for and use of PrEP among BW. Speciﬁcally, the intervention will: 1) encourage BW to access and use PrEP; and 2) increase HCP willingness to prescribe and refer PrEP to BW. Our team will explore two aims: 1) inform and develop health messages for Project ROLE with 2023 ﬁndings from focus groups with PrEP-eligible BW and key informant interviews with HCPs providing care to BW, and 2) assess the feasibility, acceptability, and preliminary impact of Project ROLE in two real-world settings with a pilot randomized controlled trial (RCT) and a social media campaign.

Aim 1: A qualitative study using focus groups with Black women and key informant interviews with healthcare providers. (Will not be included in the clinical trial.)

Aim 2a: Pilot randomized controlled trial of a behavioral intervention with both Black women and healthcare providers.

Aim 2b: Social media marketing campaign to reach and engage Black women and healthcare providers in health communication about PrEP. (Will not be included in the clinical trial.)

The proposed research is signiﬁcant because it will connect Black women to PrEP while increasing healthcare providers willingness to prescribe and refer PrEP to them using a health communication strategy that can guide the development of subsequent vlog-based interventions to address the national EHE plan.

ELIGIBILITY:
Selection criteria for participation in pilot RCT.

Eligible participants in the category for Black Women (BW) must:

1. be a woman
2. be 18 years of age
3. have been sexually active with a man within the past 6 months
4. be fluent in English
5. have a phone or internet access

Eligible participants (i.e. PrEP-eligible BW) must not:

1. be unable to provide informed consent/assent for participation (i.e., have severe cognitive impairment hat would interfere with their ability to consent or understand study procedures)
2. have psychological distress that would prohibit them from participating in the study
3. be unable or unwilling to meet study requirements
4. be ineligible for PrEP
5. received a prescription for PrEP within 12 months6)be unable to fill out the evaluation independently

Eligible participants in the HCP category must:

1. be a credentialed HCP in Texas with privileges to prescribe and/or refer PrEP
2. BW must be a part of their patient pool at the clinical setting where they practice clinically
3. be fluent in English
4. have a phone or internet access
5. Live and/or practice medicine within a 60-mile radius of Houston/Harris County

Eligible HCP must not:

1. be unable to provide informed consent for participation (e.g. have severe cognitive impairment that would interfere with their ability to consent, or ability to understand study procedures
2. have psychological distress that would prohibit them from participating in the study
3. be unable or unwilling to meet study requirements
4. be unwilling to offer PrEP to BW patients
5. have prescribed or referred PrEP to BW within the last 12 months

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants in the category for Black Women (BW) must be a woman.
Enrollment: 78 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-08-02 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with increased willingness to access or use PrEP | baseline and day of enrollment and baseline, 1-month, 3-month, and 6-month
  To assess whether participation in Project ROLE versus usual care will increase the willingness of Black women to access and/or use PrEP
Number of healthcare providers increased willingness to prescribe and/or refer PrEP | baseline and day of enrollment and baseline, 1-month, 3-month, and 6-month
  To assess whether participation in Project ROLE versus usual care will increase the willingness of healthcare providers to prescribe and/or refer PrEP to Black women

SECONDARY OUTCOMES:
Number of Black Women started to use of PrEP | 1- month, 3-months, and 6-months follow-up visits
  To assess whether Black women started to use PrEP.
Number of PrEP prescriptions or referrals by healthcare providers | 1- month, 3-months, and 6-months follow-up visits
  Using the clinical notes of electronic clinical records at participating CHCs.
PrEP adherence among those who initiated PrEP | 3-months and 6-months follow-up visits
  Assess, using a urine drug screen, whether Black women who initiated PrEP adhered to the PrEP regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Mandy Hill, DrPH,MPH,HIVPCP, Principal Investigator — University of Texas Medical Branch, Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No